CLINICAL TRIAL: NCT02556944
Title: Mix and Match Study of Two Multifocal Intraocular Lens With Different Add Power
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: tae-young chung (Other)
Responsible Party: Sponsor-Investigator, tae-young chung, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-02-001-009
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Presbyopia
Keywords: Depth of focus
MeSH Terms: conditions — Presbyopia | interventions — Phacoemulsification; Multifocal Intraocular Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mix and matched patients (Experimental): Mix and matched patients will get phacoemulsification with multifocal intraocular lens implantation with two different add power (+2.75 diopters (D) or +3.25 D, respectively) in each eye of a patient, contralaterally.
  Interventions: Device: Phacoemulsification with multifocal intraocular lens

INTERVENTIONS:
Device: Phacoemulsification with multifocal intraocular lens — Phacoemulsification and implantation of a multifocal intraocular lens (IOL) with two different add power (+2.75 diopters (D) or +3.25 D, respectively) in each eye of a patient, contralaterally. They're called mix and matched patients.

SUMMARY:
To assess postsurgical visual acuity (distant, intermediate, near), refractive errors, contrast sensitivity, visual function and patient satisfaction after implantation of multifocal IOLs of different add power contralaterally.

DETAILED DESCRIPTION:
Multifocal intraocular lens (MIOL) is considered a prevailing alternative to restore the functional vision from far to near independent of glasses. Many clinical studies on diffractive MIOLs, refractive MIOLs, or hybrid MIOLs in enhancing quality of vision showed promising outcomes. Several studies have confirmed the satisfactory visual outcomes of Tecnis MIOL with +4.00 D add power. The purpose of study is to assess the visual performance after cataract surgery with bilateral implantation of multifocal IOL with two different add power (+2.75 D or +3.25 D) in one patient.

ELIGIBILITY:
Inclusion Criteria:

* • Age-related cataract

  * Adult at the age of 21 or older at the time of the pre-operative examination and willing to have surgery on their 2nd eye within 7-28 days of their 1st eye.
  * A patient has the visual potential of 20/25 or better in each eye after cataract removal and IOL implantation.
  * A patient with preoperative corneal astigmatism from IOL Master less than 1 diopters
  * Written informed consent to surgery and participation in the study

Exclusion Criteria:

* • Pregnant woman and lactating woman

  * A patient with history of retinal disease
  * A patient with history of ocular trauma or ocular surgery (Intraocular surgery, refractive surgery, ocular surface surgery) in either eye
  * A patient with evidence of keratoconus or significant irregular astigmatism on pre-operative topography in either eye.
  * A patient that has been wearing PMMA lenses within 6 months, gas permeable lenses within one month, or extended -wear or daily soft contact lens within 7 days of their scheduled surgery.
  * Those with other diseases that can affect capsule stability such as pseudoexoliation syndrome, glaucoma, traumatic cataract, or marfan syndrome
  * Those who are not able to read and understand the informed consent (illiterate or foreigners)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Visual acuity(Distant, intermediate, near) | 1month

SECONDARY OUTCOMES:
Visual acuity(Distant, intermediate, near) | 3month

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Chung, PhD, Study Chair — Samsung Medical Center

REFERENCES:
- [Derived] Yang CM, Lim DH, Hwang S, Hyun J, Chung TY. Prospective study of bilateral mix-and-match implantation of diffractive multifocal intraocular lenses in Koreans. BMC Ophthalmol. 2018 Mar 7;18(1):73. doi: 10.1186/s12886-018-0735-0. PMID 29514611